CLINICAL TRIAL: NCT01133249
Title: Total Hip Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heekin Orthopedic Research Institute (Other)
Collaborators: Stryker Orthopaedics (Industry); DePuy Orthopaedics (Industry); Restor3D (Industry)
Responsible Party: Principal Investigator, R. David Heekin, MD, R. David Heekin, M.D., Heekin Orthopedic Research Institute
Other Study IDs: 05-09-01
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis
Keywords: total hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total hip: all consented patients receiving total hip arthroplasty

SUMMARY:
Objective

Describe the clinical and demographic characteristics of patients who undergo hip arthroplasty and document post operative outcomes.

Examine the relationship between processes of care, hospital and surgeon associated outcomes

Provide expanded data to characterize existing and evolving practice patterns, delivery of care, and resource utilization in the management of knee arthroplasty patients.

Analyze and design ancillary studies to address unanswered questions.

Disseminate findings through publication in peer-reviewed scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires total hip Arthroplasty
* Patient has signed IRB approved informed consent

Exclusion Criteria:

* Less than 21 years of age
* Patient is a prisoner

Ages: 21 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: All total hip replacements
  Selection: Males and non-pregnant females over the age of 21
Sampling Method: Non-Probability Sample
Enrollment: 942 (Estimated)
Dates: Start 2005-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 2 weeks, 6 weeks, 3 months, 6 months, 1, 2, 5, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Heekin, MD, Principal Investigator — Heekin Orthopedic Specialists
Locations (1):
- Heekin Orthopedic Specialists, Jacksonville, Florida, United States